CLINICAL TRIAL: NCT02293070
Title: One More Magnetic Resonance Imaging
Acronym: OMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-104
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Repeat Cardiac MRI Post Cryoablation (Experimental): All subjects in this study receive a follow up delayed enhanced cardiac MRI 2-6 weeks after they undergo a cryoablation procedure.
  Interventions: Other: Delayed Enhanced Cardiac Magnetic Resonance Imaging; Procedure: Cryoablation

INTERVENTIONS:
Other: Delayed Enhanced Cardiac Magnetic Resonance Imaging — Subjects in this study get a Delayed Enhanced Cardiac Magnetic Resonance Imaging 2-6 weeks after they undergo cryoablation for atrial fibrillation. This MRI is compared to the pre-procedure cardiac MRI to determine if it possible to visualize the cryoablation lesions.
  Other Names: Delayed Enhanced Cardiac MRI
Procedure: Cryoablation — All subjects in this study undergo a cryoballoon ablation procedure to achieve pulmonary vein isolation for the purposes of treatment of atrial fibrillation
  Other Names: Cryoballoon Ablation

SUMMARY:
The objective of this study is to utilize delayed enhanced cardiac magnetic resonance imaging to assess the success of pulmonary vein isolation after cryoablation of paroxysmal atrial fibrillation. The primary hypothesis is that cardiac magnetic resonance imaging will be able to visualize changes in left atrial tissue characteristics caused by cryoablation used to treat paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in the world, affecting 1-2% of the general population and 10% of people older than 80 years old. Medical therapy is only partially effective at treatment of symptoms of atrial fibrillation and ablation procedures have been developed that offer a potential curative approach to treatment of the symptoms of atrial fibrillation. Prior to an ablation procedure, it is standard of care to perform imaging (either contrast cardiac computed tomography or cardiac magnetic resonance (CMR) imaging) to determine the size and orientation of the pulmonary veins, the presence or absence of left atrial thrombus and the size and volume of the left atrium. Cardiac magnetic resonance imaging has the advantage of high spatial resolution without additional radiation exposure. There are some additional features of CMR that make it potentially even more useful for patients undergoing an ablation procedure for treatment of atrial fibrillation. One main advantage involves the use of delayed-enhancement MRI (DE-MRI) to characterize the tissue of the left atrium to visualize the presence of absence of scars. Prior studies have demonstrated the ability of CMR to visualize radiofrequency-induced scar in the left atrial wall after atrial fibrillation ablation. These studies have postulated that CMR could be utilized to determine the success rates of atrial fibrillation ablation. However, there has been significant variability between published studies looking at CMR post radiofrequency ablation, which for many years was the only type of ablation procedure available to treat atrial fibrillation. Some studies demonstrate a correlation between DE-MRI and ablation lesions, while others do not report such a correlation. Furthermore, no study to date has been designed to examine cryoablation specifically. Cryoablation is alternative method of performing an ablation procedure that utilizes a freezing balloon to make a circumferential lesion around the atrum of the pulmonary vein, as opposed to radiofrequency ablation which uses a catheter to create the same pattern of lesions around the pulmonary vein utilizing a 4mm catheter that generates heat as a byproduct of radiofrequency energy. Using DE-MRI to analyze injury and scar after cryoablation would be a novel application of this imaging modality.

There are several reasons why lesions produced with cryoablation procedures may offer better visualization on DE-MRI as compared to radiofrequency ablation. First, the circumferential lesion generated by cryoablation is created utilizing a uniform distribution of energy in a simultaneous fashion to the entire pulmonary vein antrum. In contrast, lesions created by radiofrequency ablation are produced sequentially and each lesion has variable contact with the myocardium and therefore variable energy delivery. As a consequence, lesions created with radiofrequency ablation may not uniformly penetrate the myocardium, creating a situation whereby contiguous lesions have variable depth. This may explain the heterogeneity of scar visualization on DE-MRI in earlier studies. Furthermore, despite the advantages and accuracy of electroanatomical mapping, due to variations in tissue architecture in the pulmonary vein antrum, there may be technical challenges in ensuring truly contiguous lesions. Unfortunately, the non-contiguous nature of radiofrequency ablation lesions may not be become evident until localized tissue edema has subsided and clinical evidence of recurrent atrial fibrillation is observed several months after the procedure. Cryoablation offers a theoretical advantage in this regard by producing near uniform tissue contact as well as an ability to assess for gaps in tissue contact by injecting contrast dye under fluoroscopic visualization during the period of pulmonary vein occlusion to demonstrate areas of poor tissue contact where contrast dye escapes from the occluded pulmonary vein. Another advantage is that the cryoballoon is in contact with a greater amount of myocardium in the pulmonary vein antrum than the radiofrequency ablation catheter due to the larger surface area of the 23 or 28mm diameter cryoballoon as compared to the 3.5 or 4mm diameter radiofrequency ablation catheter. The smaller surface area of the radiofrequency ablation lesions may be missed in the delayed enhancement sequences on MRI, which are acquired at a greater slice thickness as compared with standard acquisition. Therefore, the cryoablation lesions may be more likely to be visualized, as there is a greater probability that some portion of the ablated myocardium will be present in a given imaging slice of delayed enhanced atrial myocardium. Finally, the nature of cryoablation itself may cause less inflammation in the short term in the atrial myocardium as compared to radiofrequency ablation due to the fact that the tissue is frozen and not heated. The effect of this on ability to visualize ablated tissue on DE-MRI is unknown, as none of the published studies have examined cryoablation specifically.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 80 years
* A diagnosis of symptomatic paroxysmal atrial fibrillation refractory to medical therapy and planned to undergo a cryoablation procedure.

Exclusion Criteria:

* Unable or unwilling to undergo magnetic resonance imaging (including implanted metal prosthesis, severe claustrophobia and inability to tolerate sedation)
* Previous atrial fibrillation ablation
* Patients who are not candidates for cryoablation procedure for treatment of atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Visualization of late gadolinium enhancement in the pulmonary veins on cardiac MRI | 2-6 weeks after ablation
  The signal intensity of late gadolinium enhancement in the pulmonary vein region as measured on a cardiac MRI, in comparison to the signal intensity of the blood pool

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation | 3-6 months after ablation
  Electrocardiogram recording of atrial fibrillation of at least 30 seconds in duration recorded on a 30 day event montor performed 3-6 months post ablation

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya Gupta, MD, Principal Investigator — Saint Luke's Health System
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States